CLINICAL TRIAL: NCT03014882
Title: Sperm DNA Damage in β-thalassemia Major: Is There a Role for Antioxidants?
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Alaa Youssef Ahmed, Dr, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endocrinology PECASU
Record Dates: First submitted 2017-01-06; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Endocrine Disease; Fertility Decreased Male; DNA Damage
MeSH Terms: conditions — Endocrine System Diseases | interventions — Carnitine; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Antioxidant treatment (Other)
  Interventions: Drug: L-Carnitine and N-acetyl cysteine

INTERVENTIONS:
Drug: L-Carnitine and N-acetyl cysteine

SUMMARY:
Accumulation of iron in patients with beta thalassemia major causes free radical formation which leads to damage of biological membranes. Sperm DNA damage may result from these generated antioxidants.

We aimed at investigating the current DNA damage in the sperms of adult patients with beta thalassemia major and the effect generated by giving antioxidant treatment for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Pubertal patients with beta thalassemia major

Exclusion Criteria:

* Associated endcrinopathy

Min Age: 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
DNA fragmentation index | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Heba H Elsedfy, Professor, Principal Investigator — Ain Shams University
Locations (3):
- Egypt (3):
  - Ain Shams University Hospitals, Cairo Governorate, Cairo Governorate
  - Ain Shams University, Cairo
  - Ain Shams University, Cairo Governorate

IPD SHARING:
Plan to Share IPD: Undecided